CLINICAL TRIAL: NCT01469715
Title: A Clinical Study of the Warm-Up, Accuracy, and Lag Performance of a Glucose Blinding Protein-Based Continuous Glucose Monitor (GBP CGM)
Brief Title: A Clinical Study of the Performance of a Glucose Blinding Protein-Based Continuous Glucose Monitor (GBP CGM)
Acronym: SMA002
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); Becton, Dickinson and Company (Industry)
Responsible Party: Principal Investigator, Stacey Anderson, Assistant Professor, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 15696
Record Dates: First submitted 2011-11-07; First posted 2011-11-10 (Estimated); Results first posted 2015-07-31 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Continuous Glucose Monitor
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GBP-CGM (Experimental): All participants will wear one active GBP-CGM and one inactive GBP-CGM
  Interventions: Device: GBP CGM

INTERVENTIONS:
Device: GBP CGM — Visit 1: Screening visit to determine if subject qualifies for the study. Visit 2: Inpatient admission requiring a 25.5-hour hospital stay. Each subject will wear one active & one mock device simultaneously during hyperglycemic & hypoglycemic challenge conditions to observe a wide range of glucose values. Visit 3 & 4: Subjects will return to the research center approximately 24 & 48 hours after sensor removal, respectively, for evaluation of the postimplantation sensor site. Visit 5: Subjects will return to the research center approximately 28 days post inpatient admission. Blood samples for future testing of GBP and polyethylene Glycol neutralizing antibodies will be taken at Visit 1 & 5.
  Other Names: Glucose binding protein-based continuous glucose monitor

SUMMARY:
The purpose of this study is to assess the accuracy of the Becton Dickenson (BD) Technologies Glucose Binding Protein-Based Continuous Glucose Monitor (GBP CGM) in patients with Type 1 diabetes during low (goal glucose 55 mg/dL), normal (80-140 mg/dL) and high (>180mg/dL) glucose levels over a 24 hour period. This will be achieved by monitoring blood sugar levels when a regular dinner meal is given, when a liquid breakfast meal (BOOST Original containing 41 grams Carbohydrates (CHO), 4 grams fat, 10 grams protein) is given, when subcutaneous insulin is dosed to induce hypoglycemia to a goal of 55 mg/dL, and when a regular lunch meal is given. A Continuous Glucose Monitor (CGM) is an electronic device that measures and displays blood sugar (glucose) levels in the body throughout the day and night. The method being used to detect blood sugar in the investigational Glucose Binding Protein-Based Continuous Glucose Monitor (GBP CGM) is different than the method that is currently in use by commercially available models.

Some sensors cannot tell the difference between glucose (sugar) and other substances such as Tylenol, aspirin or citric acid etc. Because they cannot tell the difference, they may give false readings. The GBP CGM is made to only recognize glucose in the body rather than other substances (e.g., Tylenol, aspirin, citric acid, etc.). As a result, the investigators expect the new GBP CGM to be more accurate at detecting low blood sugar levels than the current devices.

DETAILED DESCRIPTION:
Development of accurate continuous glucose monitoring devices is critically important for the maintenance of strict glycemic control without increasing the risk for hypoglycemia and for the successful implementation of an artificial pancreas. Glucose binding protein-based (GBP) continuous glucose monitors offer several potential advantages over commercially available glucose oxidase based sensors. Unlike glucose oxidase based sensors, GBP sensors do not require establishment of an equilibrium reduction/oxidation reaction and are not as susceptible to interference from other compounds because they are engineered to recognize only glucose. As a result, GBP-based glucose sensors are exceptionally accurate at low blood glucose levels and have a faster warm-up time than glucose oxidase based systems. The principal idea of this proposal is to evaluate the accuracy and performance of a second generation glucose binding protein-based continuous glucose monitor (GBP CGM) developed by BD Technologies in subjects with type 1 diabetes, with emphasis on warm-up period after insertion, accuracy in hypoglycemic and hyperglycemic ranges, and lag time over a 24 hour period of sensor use. In order to accomplish this, the investigators will conduct a clinical trial consisting of 25.5-hour studies involving 15 subjects, each wearing one active and one mock (no GBP) device simultaneously during meals and induced hypoglycemia to observe a wide range of glucose values. The investigators envision that the glucose binding protein-based continuous glucose monitor will demonstrate minimal warm-up time after insertion, overall accuracy comparable to commercial glucose oxidase sensors with excellent performance in the hypoglycemic range and a nominal lag time to sensing a change in blood glucose.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 1 diabetes mellitus for ≥1 year. For an individual to be enrolled at least one criterion from each list must be met.
* Criteria for documented hyperglycemia (at least 1 must be met):

  1. Fasting glucose ≥126 mg/dL - confirmed
  2. Two-hour oral Glucose Tolerance Tests (OGTT) glucose ≥200 mg/dL - confirmed
  3. HbA1c ≥6.5% documented - confirmed
  4. Random glucose ≥200 mg/dL with symptoms
  5. No data at diagnosis is available but the participant has a convincing history of hyperglycemia consistent with diabetes
* Criteria for requiring insulin at diagnosis (1 must be met):

  1. Participant required insulin at diagnosis and continually thereafter
  2. Participant did not start insulin at diagnosis but upon investigator review likely needed insulin (significant hyperglycemia that did not respond to oral agents) and did require insulin eventually and used continually
  3. Participant did not start insulin at diagnosis but continued to be hyperglycemic, had positive islet cell antibodies - consistent with latent autoimmune diabetes in adults (LADA) and did require insulin eventually and used continually
* Use of an insulin pump to treat his or her diabetes for at least six months prior to the study.
* Actively using a bolus calculator function with the current insulin pump with pre-defined parameters for glucose goal(s), carbohydrate ratio(s), and insulin sensitivity factor(s).
* Signed informed consent
* Age ≥21 and <65 years old
* Body mass index between 19 and 30 kg/m2, inclusive
* HbA1c ≤11%

Exclusion Criteria:

* Uncontrolled arterial hypertension (diastolic blood pressure >90 mm Hg and/or systolic blood pressure >160 mm Hg)
* Impaired hepatic function measured as alanine aminotransferase or aspartate aminotransferase ≥three times the upper reference limit
* Impaired renal function measured as creatinine >1.2 times above the upper limit of normal
* Diabetic ketoacidosis in the past 6 months
* Severe hypoglycemia resulting in a seizure or loss of consciousness in the 12 months prior to enrollment
* Conditions which may increase the risk of induced hypoglycemia such as known coronary artery disease, congestive heart failure, history of any cardiac disorder or arrhythmia, history of a cerebrovascular event, history of migraines, seizure disorder, syncope, adrenal insufficiency, or neurological disease.
* Current use of medications containing >4000 mg acetaminophen per day.
* Current use of L-Monoamine oxidases (MAO) inhibitors.
* Known microvascular (diabetic) complications (other than diabetic non-proliferative retinopathy),such as history of laser coagulation, proliferative diabetic retinopathy, known diabetic nephropathy (other than microalbuminuria with normal creatinine) or neuropathy requiring treatment
* Known allergy to eggs
* Pregnancy, breast-feeding or intention of becoming pregnant
* Current or recent alcohol or drug abuse by patient history.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-11; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stacey Anderson, MD, Principal Investigator — University of Virginia, Center for Diabetes Technology
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GBP-CGM
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | GBP-CGM
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 4
Duration of Diabetes [Mean (Standard Deviation); unit: years] — Time since diagnosis of Type 1 Diabetes
  years | 22 (11)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Relative Difference (ARD)
Description: ARD=100*(G_sensor-G_reference)/G_reference
  Calculated for when patient's G_ref was Normal (70-180 mg/dl), Hyperglycemic (>180 mg/dl) and Hypoglycemic (<70 mg/dl)
  The study data includes 208 paired sensor-YSI plasma glucose readings (G_reference) for each GBP CGM sensor (G_sensor) inserted for 24 hours during hyperglycemic and hypoglycemic challenge conditions. Data pairs will permit the detailed evaluation of sensor performance parameters, including static accuracy metrics such as median and mean absolute deviations and median and mean absolute relative deviation and Point CG-EGA, as well as dynamic parameters, such as warm-up time, trend accuracy (Rate CG-EGA), and sensor lag.
Time Frame: 25.5 hours
Measure: Number; unit: percentage of error
Arm/Group | GBP-CGM
Number analyzed (Participants) | 12
percentage of error
  Overall | 19.1
  Hyperglycemia (>180mg/dl) | 14.9
  Hypoglycemia (<70mg/dl) | 21.8
  Normal (70-180mg/dl) | 20.4

ADVERSE EVENTS:
Arm/Group | GBP-CGM
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 4/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GBP-CGM (N=16)
Erythema (score=2) (Skin and subcutaneous tissue disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes